CLINICAL TRIAL: NCT06689813
Title: Effect of Vitamin D Supplementation on Severity of Stress Urinary Incontinence in Premenopausal Women With Vitamin D Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sheema Yousuf, second fellowship trainee in urogynaecology, Shalamar Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB - 597 - 8
Record Dates: First submitted 2024-11-01; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Stress Urinary Incontinence
Keywords: vitamin D; stress urinary incontinence; premenopausal; incontinence questionnaire short form
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Vitamin D; ispaghula seed

STUDY DESIGN:
Intervention Model Description: Group A was given oral vitamin D supplements Group B was given isphagula husk tablets
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Active Comparator): Group A participants received vitamin D supplements orally for 8 weeks along with pelvic floor exercises
  Interventions: Dietary Supplement: Vitamin D tablets
- Placebo group (Placebo Comparator): Group B participants received ispaghula husk tablets for 8 weeks along with pelvic floor exercises
  Interventions: Other: Ispaghula husk

INTERVENTIONS:
Dietary Supplement: Vitamin D tablets — Vitamin D supplements is thought to reduce the severity of urinary incontinence.Vitamin D supplements were given to Group A
  Arms: Vitamin D group
Other: Ispaghula husk — Ispaghula husk tablets were given to Group B participants
  Arms: Placebo group

SUMMARY:
The rationale for conducting the study is based on the fact that stress urinary incontinenc is a prevalent condition among middle age or older women and Vitamin D deficiency may have clinical effects on the pelvic floor muscles and bladder function. Therefore, the study aims to explore the potential link between vitamin D levels and SUI in women in our local population.

DETAILED DESCRIPTION:
The aging process is often associated with a gradual decline in muscle strength, including the weakening of pelvic floor muscles which are largely responsible for pelvic organ support and urinary retention. Weakness of these muscles is linked with urinary incontinence, the most frequently reported symptom of pelvic floor disorders. The most common type of urinary incontinence is stress urinary incontinence (SUI), which affects about 50% of women with increase in incidence with advancing age. The prevalence of stress urinary incontinence is approximately 23.58% in Pakistani middle aged women aged 40-50.

SUI occurs during times of elevated intraabdominal pressure (e.g., sneezing, coughing, and exercise). The levator muscles are responsible for supporting pelvic organs and maintaining the closure of the urethra. Strengthening the pelvic floor muscles through exercise and training is recommended as an effective treatment for SUI. The smooth and skeletal muscles throughout the body have vitamin D receptors. The pelvic floor muscles also express Vitamin D receptors, therefore Vitamin D insufficiency has shown asignificant association with pelvic floor dysfunction. Pelvic floor dysfunction includes symptoms of fecal incontinence, urinary incontinence and pelvic organ prolapse.

This study was conducted to see the association of vitamin D supplementation with improvement in stress incontinence symptoms.

Participants will be explained that their blood will be drawn twice in the study and they need to fill questionnaires with the help of principal investigator. They will be requested to sign a consent form and they will be assured that they can withdraw from the study at any time. SUI will be assessed by completing the standard ICIQ-SF (Incontinence Questionnaire - Urinary Incontinence Short) questionnaire at baseline and Serum concentrations of 25-hydroxy vitamin D will be tested by the ELISA immunoassay as per the protocol of the manufacturer.

The pateints will be divided into two groups by randomization. Group A ( intervention group) and group B (placebo group).All the patients in both groups will be advised pelvic floor exercises which is the standard first line management for stress urinary incontinence. Each study participant will be requested for 3ml of venous blood to determine their vitamin D3 levels. The treatment group will be asked to take vitamin D3 (cholecalciferol)(50,000IU) tablets, once a week, for 8 weeks and control group will be taking placebo ( isphagol husk capsules) weekly for 8 weeks. The research participants will be unaware of the type of preparation being given to them. The principal investigator will be aware of the preparation being given (single blind study).

A telephone check will be done on weekly basis to ensure intake of medication. After 8 weeks vitamin D3 levels will be checked again and standard ICIQ-SF will be assessed at month 1, month 2, and month 3. We expect participants will be enrolled in 2 months. The baseline sample will be analysed in one batch and post intervention sample will be analysed in second batch to minimize bias. Blood will be drawn by the trained phelbotimist under aseptic conditions, The samples will be stored at -80 degree centigrade in two aliquots. One will be used for measuring vitamin D and other will be for emergency purpose if required. If not used it will be discarded as per policy of Shalamar hospital. All the tests will be done in batches using ELISA-kit measuring 25 hydroxy vitamin D as per protocol of the manufacturer. The results will be entered into patient file and research reports provided by research department. Data will be recorded in the electronic system and reports will be given to the participants on their subsequent visits or will be posted to them via whattsapp by the principal investigator.

In case of any adverse drug reaction the patient will report to the principal investigator by telephonic contact and will be managed in emergency of Shalamar Hospital. Expenses for management in emergency will be given by principal investigator. Any adverse event will be reported to the IRB committee by the principal investigator.

Scoring of the stress urinary incontinence will be done based on the questions. The score ranges between 0 to 21. 1-5 (mild), 6-12 (moderate), 13-18 (severe), 19-21 (very severe). Assessment of the improvement of symptoms will be according to the change in severity(mild, moderate, severe or very severe). If the severity decreases as explained in the proforma the treatment will be considered effective The payment of laboratory tests and supplements will be given by research grant from Shalamar medical and dental college Data will be analyzed using the Statistical Package of Social Sciences SPSS version 25.0. Quantitative variables like age, number of deliveries, weight (kg), height (cm). BMI (kg/m2), serum levels of vitamin D (ng/ml) and standard ICIQ-SF score will be presented as Mean+/-SD. Qualitative variables like the impact of the severity of urinary incontinence on life as frequency and percentages. Data will be stratified for weight and number of deliveries. Chi-square test will be used for analyzing urinary incontinence between the two groups. Paired T test will be used to compare the severity of urinary incontinence and quality of life before and after intervention. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Women age between 40-49 years
  * Women with SUI

Exclusion Criteria:

* Using hormonal medications (estrogen supplementation)

  * Undergoing urogenital-related surgery (incontinence and prolapse surgery)
  * Diabetes Mellitus
  * Participants with any disorder that interferes with vitamin D absorption, such as inflammatory bowel disease, intestinal bypass surgery, or chronic liver or kidney disease
  * Neurological disease affecting the urinary system such as multiple sclerosis, degenerative muscle disease, spinal cord injury
  * Women with urinary tract infections
  * Women taking supplements ( multivitamins or already taking vitamin D supplementation)

Ages: 40 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 86 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
to see the effect of vitamin supplementation on severity of urinary incontinence | 0,4,8 and 12 weeks of treatment
  Scoring of the stress urinary incontinence was done based on the International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form Questionnaire. Severity of SUI was based on these scores, 1-5 (mild), 6-12 (moderate), 13-18 (severe), 19-21 (very severe).

SECONDARY OUTCOMES:
Impact on qulaity of life | 0,4,8 and 12 weeks of treatment
  The ICIQ-SF questionnaire(International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form) included six questions that examined the SUI condition over the past 4 weeks. Items 1 and 2 referred to demographic variables, while item 3 for urinary incontinence frequency. Item 4 measured leakage volume and item 5 evaluated impact on quality of life. Scoring of the stress urinary incontinence was done based on the Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Institute of Health Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided